CLINICAL TRIAL: NCT05207592
Title: Translation of Foot and Ankle Disability Index Into Local Urdu Language of Pakistan: A Reliability and Validity Study
Brief Title: Urdu Version of Foot and Ankle Disability Index: A Reliability and Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00267
Record Dates: First submitted 2022-01-24; First posted 2022-01-26 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Plantar Fascitis
Keywords: Foot and Ankle Disability Index; Plantar Fascitis; Cultural adaptation; Validity; Urdu Version; Reliability

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research is to translate Foot and Ankle Disability Index in Urdu and determine the validity and reliability in patients with plantar fasciitis and correlate IT with Quality of Life Short Form-36 and the Visual Analog Scale.

DETAILED DESCRIPTION:
As per recommendation of the English Version of Foot and Ankle Disability Index will be translated and culturally adapted. Foot and Ankle Disability Index along with its correlation scales will be distributed in the seventy plantar fasciitis population that will be selected according to inclusion exclusion criteria and through convenience sampling technique. To check the inter and intra observer reliability of Foot and Ankle Disability Index, Short Form-36 to measure the quality of life and Visual Analog Scale to measure pain will be filled by participants.

ELIGIBILITY:
Inclusion Criteria:

* Inability to achieve 20 degrees of active dorsiflexion
* Heel pain
* Mid foot pain
* Heal swelling
* Mid foot swelling
* Achilles' tendon tightness diagnosed on the base of Windlass test

Exclusion Criteria:

* Recent foot injury
* Fracture
* Infections
* Surgical procedures
* Tendon injury
* Hypermobility
* Neuromuscular disorders
* Impaired sensation
* Open sores
* Skin disease
* Active deep vein thrombosis or thrombophlebitis
* Bruises
* Varicose veins
* Burn Scars

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The participant included in this study will be the patients of plantar fasciitis including both genders.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Foot and Ankle Disability Index | 1st day
  The Foot and Ankle Disability Index is a 34-item questionnaire with two subscales: the Foot and Ankle Disability Index and the Foot and Ankle Disability Index Sport. Foot and Ankle Disability Index has 26 items, whereas Foot and Ankle Disability Index Sport has 8. The Foot and Ankle Disability Index includes four pain-related measures and twenty-two activity-related items. The Foot and Ankle Disability Index Sport kit includes eight activities-related products. It evaluates harder activities that are necessary in sports. The Foot and Ankle Disability Index Sport is distinct in that it is a population-specific subscale created specifically for athletes.
36-Item Short Form Survey | 1st day
  The 36-Item Short Form Survey is a popular, well-researched self-reported health assessment. It is based on the Medical Outcomes Study, which consists of 36 questions covering eight areas of health:, Limitations in physical activities due to health issues, Limitations in social activities due to physical or mental issues, Restrictions in normal role activities due to physical health issues, Bodily discomfort, General mental health (psychological distress and well-being), Restrictions in regular role activities due to emotional issues, Vitality (energy and tiredness), General health perceptions. The 36-Item Short Form Survey is frequently used to assess a person's or population's quality of life.
Visual Analogue Scale | 1st day
  A Visual Analogue Scale is a measuring tool that attempts to quantify a trait or attitude that is thought to span throughout a range of values and cannot be easily quantified directly. It is frequently used in epidemiologic and clinical research to assess the severity or frequency of different symptoms. A patient's level of pain, for example, might range from none to high. From the patient's point of view, this spectrum seems continuous; their pain does not appear to have distinct leaps, as a classification of none, mild, moderate, and severe would imply. The Visual Analogue Scale was created to capture the concept of an underlying continuity.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No